CLINICAL TRIAL: NCT06140173
Title: Randomized Controlled Trial of Low-osmolar Water Soluble Contrast Agent in Management of Adhesive Small Bowel Obstruction
Brief Title: Low-osmolar Water Soluble Contrast Agent in Management of Adhesive Small Bowel Obstruction
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Savang Vadhana Memorial Hospital, Thailand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 029/2565
Record Dates: First submitted 2023-11-14; First posted 2023-11-18 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Small Bowel Adhesion; Small Bowel Obstruction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Contrast group (CG) (Experimental)
  Interventions: Procedure: Low osmolar contrast
- Traditional group (TG) (Active Comparator)
  Interventions: Procedure: Sterile water

INTERVENTIONS:
Procedure: Low osmolar contrast — 100 mL of 350 mg omnipaque will be administered via nasogastric tube
  Arms: Contrast group (CG)
Procedure: Sterile water — 100 mL of sterile water will be administered via nasogastric tube
  Arms: Traditional group (TG)

SUMMARY:
Adhesive small bowel obstruction (ASBO) is a condition that is commonly found in patients with history of abdominal surgery. The management for such condition can be controversial. In terms of conservative treatment, recent studies have shown conflicting outcomes on whether water soluble contrast would provide benefit in reducing number of patients needed for surgery. In addition, there are a limited number of literature that investigates the role of low-osmolar contrast in reducing operative need in patients diagnosed with ASBO.

The objective of this study is to compare the operative rate of patient diagnosed with ASBO between patients who were treated with low osmolar water soluble contrast (Iohexol) and patients who were treated traditionally.

DETAILED DESCRIPTION:
This study is a randomized, controlled and double-blinded study, where participants who were diagnosed with ASBO will be randomly allocated into two groups:

(i) A contrast group (CG): Patients will be treated conservatively and received Omnipaque (Iohexol) via nasogastric tube

(ii) A traditional group (TG): Patients will be treated conservatively and received sterile water via nasogastric tube

After obtaining informed consent, the patient will be administered with either 100 mL of 350 mg Omnipaque or 100 mL of sterile water via nasogastric tube. The nasogastric tube will be clamped for 1 hour and patient will be positioned with 30 degree head elevation. In the contrast group (CG), surgery is indicated when contrast failed to reach the colon. Failure of conservative treatment is considered when there are no clinical improvements after 48 hours and the patient will then be proceeded for surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are presented with clinical manifestation of small bowel obstruction due to adhesion and require radiological investigations
* Patients who has history of abdominal surgery over 30 days

Exclusion Criteria:

* Patients with clinical signs and symptoms of bowel strangulation, ischemia, perforation or peritonitis
* Patients with clinical signs and symptoms of bowel obstruction from non-adhesive causes, including malignancy, herniation, inflammatory bowel disease, Crohn's disease, and others.
* Patients who has history of allergy to water soluble contrast agent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Rate of operative intervention | At 72 hour
  Patients who developed signs of peritonitis or failed conservative treatment or no clinical improvement after 72 hours will be managed surgically